CLINICAL TRIAL: NCT00118989
Title: Phase II Double Blind Placebo-Controlled Trial of Curcuminoids' Effect on Cellular Proliferation, Apoptosis and COX-2 Expression in the Colorectal Mucosa of Subjects With Recently Resected Sporadic Adenomatous Polyps
Brief Title: Curcumin for the Chemoprevention of Colorectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not be completed due to technology problems and cost constraints
Sponsor: University of Pennsylvania (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 802193
Record Dates: First submitted 2005-07-02; First posted 2005-07-12 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Adenomatous Polyps
Keywords: Curcumin; chemoprevention; adenomatous polyps; colorectal cancer
MeSH Terms: conditions — Adenomatous Polyps; Colorectal Neoplasms | interventions — Diarylheptanoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- PLACEBO (Placebo Comparator): placebo to be taken orally via capsule form in the dose of 4 grams daily for a duration of four months
  Interventions: Dietary Supplement: Curcuminoids
- Curcuminoids C3 Complex® to be taken orally via caps (Experimental): Curcuminoids C3 Complex® or placebo to be taken orally via capsule form in the dose of 4 grams daily for a duration of four months
  Interventions: Dietary Supplement: Curcuminoids

INTERVENTIONS:
Dietary Supplement: Curcuminoids — Curcuminoids C3 Complex® or placebo to be taken orally via capsule form in the dose of 4 grams daily for a duration of four months
  Other Names: Curcuminoids C3 Complex® (Sabinsa Co.)

SUMMARY:
Specific Aims:

* To determine if curcuminoids modulate cellular proliferation as measured by proliferating cell nuclear antigen (PCNA) in the colorectal mucosa of subjects with previously resected adenomatous colonic polyps.

Hypothesis: Curcuminoids decrease cellular proliferation in the colorectal mucosa of subjects with previously resected sporadic adenomatous colonic polyps.

* To determine if curcuminoids modulate apoptosis, as measured by TUNEL assay, in the colorectal mucosa of subjects with previously resected adenomatous colonic polyps.

Hypothesis: Curcuminoids increase apoptosis in colorectal mucosa of subjects with previously resected sporadic adenomatous colonic polyps.

* To determine if curcuminoids modulate COX-2 expression as measured by immunohistochemical assays in subjects with previously resected adenomatous colonic polyps

Hypothesis: Curcuminoids decrease colorectal mucosa COX-2 expression in subjects with previously resected sporadic adenomatous colonic polyps.

* To determine if curcuminoids modulate COX-2 activity as measured by urinary eicosanoids

Hypothesis: Curcuminoids decrease concentrations of urinary eicosanoids.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* A diagnosis for colon/rectal polyp resection, polypectomy
* Subjects must be able to have the capacity and must be willing to provide informed consent
* Premenopausal women must be surgically incapable of childbearing or be using a medically acceptable method of contraception (oral contraceptives, diaphragms, condoms with spermicide, IUD, progesterone injection or implant) throughout the entire length of the study
* Men should wear condoms during the duration of the study given the unknown effects of curcumin on sperm viability, fertility

Exclusion Criteria:

* Previous or current history of colorectal cancer
* Previous history of Familial Polyposis Syndromes
* Previous history of inflammatory bowel disease
* Previous surgery of the large bowel
* Liver disease defined as AST and ALT>3x upper limit of normal
* Known history of gallstones, biliary colic or serum bilirubin >2.0
* Cardiac disease including myocardial infarction, congestive heart failure, arrhythmia
* Renal disease defined as creatinine >1.5
* Hematopoietic disease defined as WBC<4000, platelet count <100,000, hemoglobin<10.0 or coagulation or bleeding disorder
* Significantly impaired gastrointestinal function or absorption
* Peptic ulcer disease
* Active infection including viral, bacterial, atypical or fungal infections of any organ system including HIV
* Previous history of allergy to turmeric, Indian curries, aspirin or NSAIDs
* Pregnant or lactating women
* Dementia or other neurologic or psychiatric disease which may impede the ability to follow the protocol
* Inability to swallow pills
* Prior or concurrent therapy with any herbal or dietary supplement containing curcuminoids
* Concurrent use of anticoagulants or antiplatelets including warfarin, clopidogrel
* Prior or concurrent use of colorectal cancer chemopreventive agents including herbals: Sulindac or other NSAIDs, aspirin, COX-2 inhibitors, 5-aminosalicylate, folate, calcium, or their use within 14 days of enrollment
* Concurrent use of immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-07; Primary Completion 2010-09 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Cellular proliferation and apoptosis in the colonic mucosa | 4 months

SECONDARY OUTCOMES:
COX-2 expression and activity | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen E Guerra, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States